CLINICAL TRIAL: NCT04013126
Title: Endothelial Dysfunction Among Woman With Endometriosis After Surgical Treatment
Brief Title: Endothelial Dysfunction Among Woman With Endometriosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Eyal Rom, MD, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0100-18-emc
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: 2 groups (treatment, control) each group is evaluated pre and post-surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- endometriosis (Experimental): Women who undergoing surgery for removal of endometriosis implants
  Interventions: Diagnostic Test: • Endothelial function using ENDOPAT system
- non-endometriosis (Active Comparator): Women who undergoing surgery for removal of benign masses in the pelvis
  Interventions: Diagnostic Test: • Endothelial function using ENDOPAT system

INTERVENTIONS:
Diagnostic Test: • Endothelial function using ENDOPAT system — All of the participants will follow an non-invasive test for endothelial function using ENDOPAT 2000 device before surgery. A consecutive assessment will be held 6 weeks and 2 years post-surgery, using the same method.

SUMMARY:
Endometriosis is a chronic disease defined as an ectopic endometrial tissue outside the, and associated with chronic inflammatory state and increased risk of atherosclerosis.

Endothelial dysfunction plays an important and elementary role in the development of atherosclerosis.

There are number of non-invasive tests for evaluating the endothelial function. One of them is FMD - "Flow Mediated Dilatation". Clinical studies proved the efficacy of this method in predicting cardio-vascular events in patients with established heart disease and also as an independent risk factor, better than the traditional ones.

An alternative method, developed in recent years, is evaluation of peripheral blood vessels tone - "Peripheral Arterial Tonometry" - (PAT). It evaluates the pulsatile blood volume of the blood vessels in the fingertips during reactive hyperemia. The obtained value "reactive hyperemic index" (RHI) correlates well with FMD as well with coronary arteries endothelial dysfunction.

it well suited as a clinical tool or as a test for a large-scale clinical study.

Endothelial dysfunction has been demonstrated among woman with endometriosis. After surgical removal of endometrial implants there was a substantial improvement in the endothelial function, by imaging (using FMD) and by inflammatory markers

In this study the investigators will follow the endothelial function among women undergoing endometrial implants surgical removal, before and after the surgery, using PAT technology (ENDOPAT system). Inflammatory markers and quality of life parameters will also be evaluated.

The follow-up will include one meeting 6 weeks after the procedure The investigators expect an improvement in the endothelial function among women who had endometriosis implants removal.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease defined as an ectopic endometrial tissue outside the uterus, mostly in the pelvis. It is related to major morbidity and infertility. It is also associated with chronic inflammatory state and increased risk of atherosclerosis.

Endothelial dysfunction plays an important and elementary role in the development of atherosclerosis.

There are number of non-invasive tests for evaluating the endothelial function. One of them is FMD - "Flow Mediated Dilatation". It refers to dilation (widening) of an artery when blood flow increases in that artery after An intentional block of the blood flow. Clinical studies proved the efficacy of this method in predicting cardio-vascular events in patients with established heart disease and also as an independent risk factor, better than the traditional ones.

An alternative method, developed in recent years, is evaluation of peripheral blood vessels tone - "Peripheral Arterial Tonometry" - (PAT). It evaluates the pulsatile blood volume of the blood vessels in the fingertips during reactive hyperemia. The obtained value "reactive hyperemic index" (RHI) correlates well with FMD as well with coronary arteries endothelial dysfunction.

The test is performed by attaching two sensors to the patient's fingertips. Using this method requires short training interval, completely user-independent and the accepted result is a quantitive index. Because it takes only 15 minute to complete the test it well suited as a clinical tool or as a test for a large-scale clinical study.

Endothelial dysfunction has been demonstrated among woman with endometriosis. After surgical removal of endometrial implants there was a substantial improvement in the endothelial function, by imaging (using FMD) and by inflammatory markers, so no difference was shown between them and healthy women, 2 years thereafter.

In a large meta-analysis, evaluating 5,547 patients, every 1% improvement in the FMD scale resulted in a 13% decrease in the rate of cardio-vascular events.

In a meta-analysis evaluating 5,547 patients a 13% reduction in the risk to cardio-vascular events was demonstrated for every 1% improvement in the FMD score.

In this study the investigators will follow the endothelial function among women undergoing endometrial implants surgical removal, before and after the surgery, using PAT technology (ENDOPAT system). Inflammatory markers and quality of life parameters will also be evaluated.

The follow-up will include one meeting 6 weeks after the procedure the investigators expect an improvement in the endothelial function among women who had endometriosis implants removal.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergoing surgery for removal of endometriosis implants

Exclusion Criteria:

* Women under 18 or above 60 years of age
* Women with known vascular disease
* Women with chronic disease which effect the endothelial function (Diabetes mellitus, Hypertension, Obesity (Defined as BMI≥30), Atherosclerosis, Kidney disease, Collagen disease, Chronic inflammatory disease, and Etc.
* History of Cardio-vascular event or venous thromboembolism (VTE)
* Smoking
* Pregnant women or gave birth in the past 3 months

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline endothelial function at 6 weeks | before and 6 weeks after surgery
  RHI index - "Reactive Hyperemia Index"
Change from baseline inflammatory markers at 6 weeks | before and 6 weeks after surgery
  C-reactive protein

SECONDARY OUTCOMES:
Change from baseline pain score at 6 weeks | before and 6 weeks after surgery
  visual analog scale (VAS)- scale for patient self-reporting of pain. 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, 7-10 represents severe pain). a lower pain level 6 weeks after surgery is a better outcome
Change from baseline quality of life score at 6 weeks | before and 6 weeks after surgery
  The Short Form (SF-36) Health Survey is a 36-item, patient-reported survey of patient health.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. a higher score 6 weeks after surgery is a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Rom, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel